CLINICAL TRIAL: NCT01851655
Title: The Effect of Plyometric Exercise Intensity on Function & Articular Cartilage Metabolism After ACL Reconstruction
Brief Title: Anterior Cruciate Ligament Reconstruction and Plyometric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: NFL Charities (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-2008
Record Dates: First submitted 2013-04-25; First posted 2013-05-10 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: rehabilitation; plyometric
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plyometric Exercise - High intensity (Experimental): The exercises should produce a higher peak vertical ground reaction force than those in the low group based on literature findings (e.g. single leg jumps, jumps from higher heights, higher percent effort).
  Interventions: Behavioral: Plyometric Exercise
- Plyometric Exercise - Low intensity (Active Comparator): A lower peak vertical ground reaction force will be generated in the low intensity group compared to the high intensity group based on findings in the literature (e.g. lower box heights, only two-legged jumps, lower percent effort)
  Interventions: Behavioral: Plyometric Exercise

INTERVENTIONS:
Behavioral: Plyometric Exercise — Treatment sessions include a combination of running, jumping and agility activities (plyometric exercise). Each rehabilitation session will also include an abbreviated, standardized program of lower extremity strengthening (leg press, machine squats, knee extensions; 3 sets x 10 repetitions each), flexibility (standing gastrocnemius and quadriceps stretch, hamstrings stretch in long-sitting; 2 x 30 seconds each) and proprioception (standing on foam and a tilt board; 3 x 30 seconds each).

SUMMARY:
This is a single-center, randomized, double-blind (subject/evaluator)study. Enrolled patients had anterior cruciate ligament (ACL) reconstruction and met criteria for advanced rehabilitation. The study included 8 weeks of advanced rehabilitation consisting of low- or high-intensity plyometric exercise. The objective of the study was to determine the effect of plyometric exercise intensity on knee function and knee cartilage in patients with ACL reconstruction.

DETAILED DESCRIPTION:
As part of the study, investigators will insure patients meet the criteria for advanced rehabilitation based on knee motion, pain levels and quadriceps strength.

Participants will be asked to review the informed consent and consent to the study prior to any study procedures. The study will consist of 2 testing sessions and an 8 week intervention (2 visits per week) at the UF&Shands Orthopaedics and Sports Medicine Institute. The testing sessions will include clinical measures of knee impairments, questionnaires, biomechanical analysis and functional performance testing.

ELIGIBILITY:
Inclusion Criteria:

1. time from injury to ACL reconstruction is no greater than 6 months,
2. pre-injury activity level includes participation in high-demand activities, and
3. meet the criteria for advanced rehabilitation including full active knee extension, active knee flexion within 5 degrees of the contralateral side, pain rating no greater or equal to 1/10 with activities of daily living, and involved side knee extensor strength at least 60% of the contralateral side.

Exclusion Criteria:

1. bilateral knee injury,
2. prior knee ligament injury and/or surgery,
3. concomitant other ligamentous injury > Grade I,
4. meniscal repair performed in conjunction with ACL reconstruction,
5. cartilage repair procedure performed in conjunction with ACL reconstruction,
6. complications during surgery requiring protocol modification, and
7. renal disease.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terese L Chmielewski, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

REFERENCES:
- [Derived] Chmielewski TL, George SZ, Tillman SM, Moser MW, Lentz TA, Indelicato PA, Trumble TN, Shuster JJ, Cicuttini FM, Leeuwenburgh C. Low- Versus High-Intensity Plyometric Exercise During Rehabilitation After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2016 Mar;44(3):609-17. doi: 10.1177/0363546515620583. Epub 2016 Jan 21. PMID 26797700

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 subjects were consented to the study. One subject who was enrolled in the study was found to have insufficient quadriceps strength to participate in the study during baseline testing. She was withdrawn prior to randomization. 24 subjects were randomized to the study.
Period: Overall Study
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sample size was based on the minimal detectable change in IKDC-SKF scores and from urinary CTX-II concentrations in uninjured athletes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.3 (3.8) | 20.7 (4.9) | 20.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in International Knee Documentation Committee (IKDC) Subjective Form Score.
Description: The IKDC subjective form is a measure of self-reported knee function. It includes items related to symptoms and functional activities. Scores range from 0 to 100 points, and higher scores equal higher function. Responses will be recorded on hard-copy and entered into a spreadsheet to calculate the score. The change will be computed as (post-intervention score minus pre-intervention score).
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
units on a scale | 15.5 (6.8) | 12.1 (7.5)

2. Primary Outcome: Change in Urinary Concentrations of the C-terminal Crosslinking Telopeptide of Type II Collagen (CTX-II)
Description: CTX-II is a biomarker of Type II collagen degradation. Early morning, second-void urine samples will be collected and stored. Concentrations of CTX-II will be determined with enzyme-linked immunosorbent assay and corrected for creatinine concentration, which will also be determined with enzyme-linked immunosorbent assay. Values will be log-transformed. The change in urinary CTX-II concentration will be computed as (post-intervention value minus pre-intervention value).
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: log-scale transformed value of ng/mmol
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
log-scale transformed value of ng/mmol | -0.1 (0.2) | -0.1 (0.1)

3. Secondary Outcome: Change in Vertical Jump Height.
Description: Vertical jump height will be assessed with the Vertex. The average of three trials will be recorded in cm. The change in vertical jump height will be computed as (post-intervention value minus pre-intervention value).
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
cm | 5.0 (4.7) | 2.6 (5.0)

4. Secondary Outcome: Change in the Ratio of Urinary CTXII to Serum CPII Concentrations.
Description: CTX-II is a biomarker of Type II articular cartilage degradation. Type II collagen carboxy propeptide (CPII) is a biomarker of Type II collagen synthesis. Early morning urine and blood samples will be collected pre- and post-treatment. Urinary CTX-II will be analyzed as described in Primary Outcomes. Serum CPII will be determined using enzyme-linked immunosorbent assay. Values of both biomarkers will be log-transformed, and the ratio of CTXII:CPII will be calculated. The change will be computed as (post-intervention CTXII:CPII values minus pre-intervention CTXII:CPII value).
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: log [(ng/mmol)/(ng/mL)]
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
log [(ng/mmol)/(ng/mL)] | 0.02 (0.06) | -0.01 (0.09)

5. Other Pre Specified Outcome: Change in Quadriceps Strength
Description: Knee extensor torque will be measured with an isokinetic dynamometer. The lever arm will move at 60 degrees/second. The peak torque from 5 trials will be obtained and normalized to body weight. The change will be computed as (post-intervention value minus pre-intervention value)
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: ft-lb/lb
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
ft-lb/lb | 0.13 (0.13) | 0.08 (0.26)

6. Other Pre Specified Outcome: Change in Fear of Movement/Re-injury
Description: The 11-item version of the Tampa Scale for Kinesiophobia will be used to assess kinesiophobia or fear of movement/re-injury. Scores range from 11 to 44 points, and higher scores equal higher fear of movement/re-injury. Responses will be recorded on hard-copy and entered into a spreadsheet to calculate the score. The change will be computed as (post-intervention score minus pre-intervention score).
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
units on a scale | 0.1 (4.1) | -0.2 (3.8)

7. Other Pre Specified Outcome: Change in Anterior Knee Laxity
Description: Anterior knee laxity will be assessed with a knee arthrometer and a maximum manual pull. The side-to-side difference will be recorded in mm. The change will be computed as (post-intervention difference minus pre-intervention difference).
Time Frame: Baseline (pre-intervention) to 9 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Number analyzed (Participants) | 12 | 12
mm | -0.1 (0.6) | -0.2 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were compiled as they occurred.
Arm/Group | Plyometric Exercise - High Intensity | Plyometric Exercise - Low Intensity
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plyometric Exercise - High Intensity (N=12) | Plyometric Exercise - Low Intensity (N=12)
Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject sustained injury to her surgical knee while performing an activity (skateboarding) that was not part of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No